CLINICAL TRIAL: NCT05481541
Title: The Effect of E-Mobile and Written Education on Quality of Life and Sleep After Transurethral Surgery
Brief Title: The Effect of E-Mobile and Written Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Seyma Yurtseven, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0000-0003-2378-682X
Record Dates: First submitted 2022-03-30; First posted 2022-08-01 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Quality of Life; Sleep; Education; Counseling; Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- written education group (Experimental): Experimental: The Effect of E-Mobile and Written Education on Quality of Life and Sleep in Patients with Transurethral Prostate Resection According to the randomization, preoperative training will be applied to the patients in the e-mobile training/written training group. The training will be administered by the principal researcher using the face-to-face interview technique.
  Interventions: Other: written education
- Mobile education application group (Active Comparator): Experimental: The Effect of E-Mobile and Written Education on Quality of Life and Sleep in Patients with Transurethral Prostate Resection According to the randomization, preoperative written/mobile education will be applied to the patients in the e-mobile education/written education group. The training will be given by the principal researcher using the face-to-face interview technique.
  Interventions: Other: written education
- Control (standard care) group (No Intervention): Experimental: The Effect of E-Mobile and Written Education on Quality of Life and Sleep in Patients with Transurethral Prostate Resection Routine post-operative care will be given to the control group without any intervention and data collection tools will be applied at the same time as the experimental group, twice at 30-minute intervals.

INTERVENTIONS:
Other: written education — Other names:
  Written/E-Mobile training The study was conducted as a three-group randomized controlled trial to examine the effect of written/mobile education on the quality of life and sleep of patients undergoing transurethral resection of the prostate. Written education was applied to the first group and mobile education was applied to the second group. Group 3 formed the control group.
  Other Names: E-Mobile education
  Arms: Mobile education application group; written education group

SUMMARY:
Bening's Prostate Hyperplasia (BPH), which is closely related to aging, is one of the most common diseases in the world. Although it is not a life-threatening condition, lower urinary tract symptoms (LUTS) are seen in many patients, which disrupts their daily activities, sleep patterns, and quality of life of the patients. Examination of changes in sleep and quality of life after transurethral resection of the prostate (TUR-P) in patients with LUTS due to BPH and planning training according to their needs will positively affect the lives of these patients. It is very important for nurses to provide individual training and counseling by making use of innovative technology to ensure that patients manage the surgical process in a healthy way and cope with possible complications. This thesis study was planned as a three-group randomized controlled experimental study in order to determine the effect of e-mobile training and counseling on quality of life and sleep in patients who underwent TUR-P to manage the operative process and cope with possible complications.

DETAILED DESCRIPTION:
This thesis study aims to determine the effect of e-mobile training and counseling on quality of life and sleep in patients who underwent TUR-P for BPH, to manage the operation process and to cope with possible complications, and to determine the effectiveness of the written training given to the patients, the control group and the e-mobile application designed for comparasion.

ELIGIBILITY:
Inclusion criteria:

- Being literate, not having communication, hearing and visual impairments, not having any psychiatric disorders, not having sleep apnea, using a smartphone for at least 1 year in the experimental group,

Exclusion Criteria:

-The patient's refusal to participate in the study

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Obligation of male gender due to the presence of prostate
Enrollment: 83 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
1. Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 [Time Frame: 0 days-3 month] | Time Frame:0-3 months
  Change in sleep and quality of life before and after training

CONTACTS AND LOCATIONS:
Overall Officials: Sevban Arslan, PhD, Study Chair — Cukurova Universty Faculty of Health Sciences Adana, Turkey
Locations (2):
- Turkey (Türkiye) (2):
  - Cukurova University, Adana, Eyalet/Yerleşke
  - Cukurova University, Adana

IPD SHARING:
Plan to Share IPD: No